CLINICAL TRIAL: NCT07340060
Title: Statistical Association Between Bicarbonate Levels and Death or Admission to Intensive Care Within 48 Hours in Patients Presenting to the Emergency Department
Acronym: BRAVOinED
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Other Study IDs: CHD25_0056
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Urgency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bicarbonate testing in patients admitted to the emergency department.: Bicarbonate testing in patients admitted to the emergency department.

SUMMARY:
Statistical Association Between Bicarbonate Levels and Death or Admission to Intensive Care Within 48 Hours in Patients Presenting to the Emergency Department

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient with blood ionogram performed upon admission to the emergency department
* Patient capable of understanding the protocol and not opposed to participating in the research

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This research is intended for adult patients admitted to the emergency department at CHD Vendée for whom an ionogram has been prescribed.
Sampling Method: Non-Probability Sample
Enrollment: 6500 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-01-06 (Estimated); Study Completion 2026-07-05 (Estimated)

PRIMARY OUTCOMES:
Composite criterion: -Admission to a critical care unit within 48 hours of admission to the emergency department. -Death within 48 hours of admission to the emergency department. | 48 hours
  Composite criterion:
  * Admission to a critical care unit within 48 hours of admission to the emergency department.
  * Death within 48 hours of admission to the emergency department.

CONTACTS AND LOCATIONS:
Overall Officials: COLIN Gwenhael, Principal Investigator — CHD Vendee

IPD SHARING:
Plan to Share IPD: No